CLINICAL TRIAL: NCT07029620
Title: Evaluation and Rehabilitation of Patients With Peripheral Neuropathy Using Static and Dynamic Stabilometric Platforms: NEUROSTAB
Brief Title: Peripheral Neuropathy Rehabilitation With Stabilometric Platforms (NEUROSTAB)
Acronym: NEUROSTAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEUROSTAB - PNC0000007; #PNC0000007 (Other Grant/Funding Number: NRRP "Fit4MedRob-Fit for Medical Robotics")
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-04

CONDITIONS: Rehabilitation; Balance
Keywords: Peripheral Neuropathy; Postural Control; Stabilometric Platform; Dynamic Balance; Static Balance; Rehabilitation; Neurorehabilitation; Balance Training
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Study type: interventional. Allocation: randomized Intervention model: parallel assignment (1:1) This study involves two treatment groups of patients with peripheral neuropathies and one additional non-treatment group of healthy subjects.
  The healthy control group is not part of the therapeutic comparison; rather, it is included exclusively for the purpose of evaluating the reproducibility of the stabilometric measurements recorded with the GEAMASTER platform.
  The main comparison of treatment efficacy is conducted only between the two patient groups.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The randomization process is conducted by a staff member who is not involved in either the treatment delivery or the outcome assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Instrumented Balance (GeaMaster) Training Group (Experimental): Participants in this arm are patients diagnosed with peripheral neuropathy who will undergo a structured rehabilitation program supported by the GEAMASTER stabilometric platform. The intervention involves balance training sessions during which the GEAMASTER device provides real-time postural feedback by measuring center-of-pressure shifts under both static and dynamic conditions.
  Interventions: Device: Balance and postural rehabilitation using sensor-based stabilometric platform (GEAMASTER) under static and dynamic conditions
- Active Comparator: Traditional Rehabilitation Training Group (Active Comparator): Participants in this arm are patients diagnosed with peripheral neuropathy who will undergo a structured rehabilitation program using traditional physiotherapy methods. The intervention includes balance and gait training exercises without technological support, such as weight shifting, static and dynamic balance tasks, and obstacle navigation performed on conventional surfaces.
  Interventions: Other: Conventional balance and gait rehabilitation program
- Reference Arm: Healthy Subjects Group (Other): Participants in this arm are healthy individuals with no history of neurological or balance disorders who will undergo stabilometric assessments using the GEAMASTER platform. The purpose of this arm is to establish normative data and evaluate the test-retest reliability of the device under both static and dynamic conditions.
  Interventions: Other: Stabilometric assessment in healthy volunteers

INTERVENTIONS:
Device: Balance and postural rehabilitation using sensor-based stabilometric platform (GEAMASTER) under static and dynamic conditions — This intervention consists of a structured postural rehabilitation program supported by the GEAMASTER stabilometric platform. The device provides real-time feedback on center-of-pressure shifts and enables both static and dynamic balance training through interactive visual tasks. Exercises include multi-directional weight shifting, stability control, and task-specific balance strategies. The platform integrates sensor-based tracking and allows fine-grained analysis of postural parameters, distinguishing it from conventional physiotherapy by its precision, adaptability, and real-time feedback mechanisms.
  Arms: Instrumented Balance (GeaMaster) Training Group
Other: Conventional balance and gait rehabilitation program — This intervention consists of a standardized physiotherapy program aimed at improving postural control and gait in patients with peripheral neuropathy. The rehabilitation protocol includes stretching, weight-shifting exercises, balance training on foam or unstable surfaces, and obstacle navigation. Unlike the experimental intervention, this program does not use any technological or sensor-based feedback systems. The content, frequency, and duration of the sessions are matched to those of the experimental arm to allow for comparative analysis of clinical outcomes.
  Arms: Active Comparator: Traditional Rehabilitation Training Group
Other: Stabilometric assessment in healthy volunteers — This intervention involves a non-interventional assessment of healthy adult volunteers using the GEAMASTER stabilometric platform. The objective is to generate normative data for stabilometric parameters and to assess test-retest reliability of the device under static and dynamic conditions. Participants do not undergo any rehabilitation program or therapeutic intervention. The data collected will serve as a reference for interpreting pathological findings in patients with peripheral neuropathy.
  Arms: Reference Arm: Healthy Subjects Group

SUMMARY:
The goal of this clinical trial is to learn if the GeaMaster stabilometric platform can support rehabilitation and improve balance and walking ability in adults diagnosed with peripheral neuropathy. It will also evaluate whether the platform can provide objective and reliable data that match the results of standard clinical tests. The study will explore if brain and muscle activity, recorded during movement, can indicate how much motor learning and recovery has occurred.

Peripheral neuropathies are disorders of the peripheral nerves and can have many causes, including diabetes, autoimmune diseases, toxins, or inherited conditions such as Charcot-Marie-Tooth disease. Symptoms may include reduced sensation, muscle weakness, poor reflexes, balance problems, and frequent falls. Since there are no approved drugs for many of these conditions, physical therapy is the main treatment option.

The main questions this study aims to answer are:

* Does using GeaMaster improve balance and walking better than traditional rehabilitation alone?
* Are GeaMaster's stabilometric data consistent with standard balance and gait test scores?
* Can movement-related evoked potentials be used as biomarkers to track and predict motor recovery? To answer these questions, researchers will compare two groups of patients. One group will receive traditional physiotherapy. The other group will receive the same therapy with the support of the GeaMaster platform. Both groups will follow the treatment for 4 weeks. A group of healthy volunteers will also be included for comparison.

Participants will:

* Be adults aged 18 to 80. Patients must have a diagnosis of peripheral neuropathy and a stable condition.
* Be randomly assigned to a control group (traditional rehab) or experimental group (rehab with GeaMaster).
* Visit the clinic for balance and walking tests at three time points: before treatment (T0), after 4 weeks of treatment (T1), and 1 month later (T2).
* Complete clinical tests such as the Berg Balance Scale, 6-Minute Walk Test, 10-Meter Walk Test, Tinetti Scale, and Modified Barthel Index.
* Be assessed using the GeaMaster platform for postural stability under both static and dynamic conditions.
* Undergo neurophysiological tests using EEG and EMG to record brain and muscle activity during tasks like walking, writing, or drawing.

Healthy volunteers will visit the clinic twice (5 days apart) to check how stable the GeaMaster measurements are over time.

GeaMaster is a robotic platform that uses compressed air to gently move the support surface and challenge a patient's balance. It offers different levels of difficulty and provides real-time visual feedback. Its design avoids mechanical inertia, making movements feel more natural and safe for patients of all ages.

The main outcome researchers will look for is a significant link between GeaMaster balance data and results of the Berg Balance Scale and the 10-Meter Walk Test. Other outcomes include performance on additional scales, the presence of balance improvements, risk of falling, and changes in movement-related brain signals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged between 18 and 80 years
* Patients aged between 18 and 80 years with a diagnosis of peripheral neuropathy, according to international criteria
* Patients must be at an equivalent stage of disease
* Patients must be undergoing comparable and analogous treatments
* Pharmacological treatment stability during the last 6 months

Exclusion Criteria:

* Severe comorbidity
* Presence of other neurological disorders or balance alterations due to other diseases (e.g., vestibular or cerebellar conditions)
* Pain with VAS >3 in any body region
* Orthopedic surgery within the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Correlation between sway area and sway path values and scores on the Berg Balance Scale | From baseline (T0) to one-month post-treatment follow-up (T2), approximately 8 weeks total
Correlation between sway area and sway path values and performance on the 10-Meter Walk Test | From baseline (T0) to one-month post-treatment follow-up (T2), approximately 8 weeks total

SECONDARY OUTCOMES:
Correlation between additional stabilometric parameters (static balance, dynamic balance, fall risk, and mobility) and clinical outcomes | From baseline (T0) to one-month post-treatment follow-up (T2), approximately 8 weeks total
Temporal and frequency domain analysis of movement-related cortical potentials in upper and lower limbs | From baseline (T0) to one-month post-treatment follow-up (T2), approximately 8 weeks total
Comparison of movement-related cortical activity in upper versus lower limbs to evaluate motor learning effects | From baseline (T0) to one-month post-treatment follow-up (T2), approximately 8 weeks total

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baratto L, Morasso PG, Re C, Spada G. A new look at posturographic analysis in the clinical context: sway-density versus other parameterization techniques. Motor Control. 2002 Jul;6(3):246-70. doi: 10.1123/mcj.6.3.246. PMID 12122219
- [Background] Scoppa F, Capra R, Gallamini M, Shiffer R. Clinical stabilometry standardization: basic definitions--acquisition interval--sampling frequency. Gait Posture. 2013 Feb;37(2):290-2. doi: 10.1016/j.gaitpost.2012.07.009. Epub 2012 Aug 11. PMID 22889928
- [Background] Wright DJ, Holmes PS, Smith D. Using the movement-related cortical potential to study motor skill learning. J Mot Behav. 2011;43(3):193-201. doi: 10.1080/00222895.2011.557751. PMID 21462065
- [Background] Shibasaki H. Cortical activities associated with voluntary movements and involuntary movements. Clin Neurophysiol. 2012 Feb;123(2):229-43. doi: 10.1016/j.clinph.2011.07.042. Epub 2011 Sep 8. PMID 21906995
- [Background] Prada V, Mori L, Accogli S, Rivarola M, Schizzi S, Hamedani M, Schenone A. Testing overwork weakness in Charcot-Marie-tooth disease: Is it true or false? J Peripher Nerv Syst. 2018 Jun;23(2):124-128. doi: 10.1111/jns.12270. Epub 2018 May 7. PMID 29693294
- [Background] Gess B, Baets J, De Jonghe P, Reilly MM, Pareyson D, Young P. Ascorbic acid for the treatment of Charcot-Marie-Tooth disease. Cochrane Database Syst Rev. 2015 Dec 11;2015(12):CD011952. doi: 10.1002/14651858.CD011952. PMID 26662471
- [Background] Rose KJ, Hiller CE, Mandarakas M, Raymond J, Refshauge K, Burns J. Correlates of functional ankle instability in children and adolescents with Charcot-Marie-Tooth disease. J Foot Ankle Res. 2015 Nov 5;8:61. doi: 10.1186/s13047-015-0118-1. eCollection 2015. PMID 26543504
- [Background] Pareyson D, Scaioli V, Laura M. Clinical and electrophysiological aspects of Charcot-Marie-Tooth disease. Neuromolecular Med. 2006;8(1-2):3-22. doi: 10.1385/nmm:8:1-2:3. PMID 16775364
- [Background] Eggermann K, Gess B, Hausler M, Weis J, Hahn A, Kurth I. Hereditary Neuropathies. Dtsch Arztebl Int. 2018 Feb 9;115(6):91-97. doi: 10.3238/arztebl.2018.0091. PMID 29478438
- [Background] Mathis S, Magy L, Le Masson G, Richard L, Soulages A, Sole G, Duval F, Ghorab K, Vallat JM, Duchesne M. Value of nerve biopsy in the management of peripheral neuropathies. Expert Rev Neurother. 2018 Jul;18(7):589-602. doi: 10.1080/14737175.2018.1489240. Epub 2018 Jun 25. PMID 29923431